CLINICAL TRIAL: NCT04756167
Title: The Effect of Myofascial Relaxation on Pain, Functionality and Quality of Life in Individuals With Adhesive Capsulitis: A Randomized Controlled Single-Blind Study
Brief Title: Effect of Myofascial Relaxation on Individuals With Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Kübra TAPAN, Physical therapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1508796
Record Dates: First submitted 2021-02-01; First posted 2021-02-16 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Adhesive Capsulitis
Keywords: muscle relaxation; quality of life; range of motion; shoulder pain; sleep
MeSH Terms: conditions — Bursitis; Shoulder Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: The individuals are randomly allocated into conventional and myofascial release groups
Who Masked: Outcomes Assessor
Masking Description: The researcher who will make the measurements will not know the treatment groups of the individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Group (Active Comparator): The treatment of 21 individuals in the conventional group will be done by the researcher. Among the conservative treatment methods, hot pack(15 minutes) around the glenohumeral joint, conventional TENS(15 minutes) for painful points, ultrasound(1.5 watt / cm² power, 5 minutes) and exercise(passive and active range of motion) approaches will be applied. Individuals will be asked to come to the center where the research will be conducted for a total of fifteen sessions for three weeks, five times a week.
  Interventions: Other: Conventional Treatment
- Myofascial Release Group (Active Comparator): Treatment of 21 individuals in the Myofascial Release group will be done by the researcher. Among the conservative treatment methods, hot pack(15 minutes) around the glenohumeral joint, conventional TENS(15 minutes) for painful points, ultrasound(1.5 watt / cm² power, 5 minutes),exercise(passive and active range of motion) and myofascial release to subscapularis and serratus anterior muscles approaches will be applied. Individuals will be asked to come to the center where the research will be conducted for a total of fifteen sessions for three weeks, five times a week. Myofascial release will be done in the first five sessions of treatment programs.
  Interventions: Other: Myofascial Release Treatment

INTERVENTIONS:
Other: Conventional Treatment — Hotpack, TENS, ultrasound and exercise
  Arms: Conventional Group
Other: Myofascial Release Treatment — Hotpack, TENS, ultrasound, exercise and myofascial release therapy for subscapularis and serratus anterior muscles
  Arms: Myofascial Release Group

SUMMARY:
In the study, the investigators aimed to investigate the effects of myofascial release method on pain, functionality and quality of life in individuals with adhesive capsulitis. 42 individuals willing to participate in the study will be included. Participants will be randomly divided into two groups, the conventional group and the myofascial release group. Evaluations will be made by another physiotherapist with a single eye blindness. Hotpack, TENS, ultrasound and exercise will be applied jointly to both groups in the study. In addition to the myofascial release group, myofascial release will be applied on the subscapularis and serratus anterior muscles. Individuals will be asked to come to the center where the research will be conducted for a total of fifteen sessions for three weeks, five times a week. Myofascial release will be done in the first five sessions of treatment programs. Participants' pain before the first treatment, at the end of the 5th treatment and after the 15th treatment with Visual Analogue Scale (VAS), shoulder joint range of motion (ROM) with Goniometer, upper extremity functionality level Arm, Shoulder and Hand Problems Questionnaire (DASH) specific shoulder pain and functions will be evaluated with the Shoulder Pain and Disability Index (SPADI), sleep quality with Pittsburgh Sleep Quality Index (PSQI), and quality of life with Short Form-36 (SF-36). Statistical analysis to be used in the investigators study will be made with the Statistical Package for the Social Sciences 20.0 package program.

DETAILED DESCRIPTION:
Adhesive capsulitis is a shoulder pathology characterized by pain persisting for more than three months due to fibrosis and contractures in the glenohumeral joint capsule, active and passive joint motion limitation and functional insufficiency. Although there are many factors that trigger this pathology, also known as frozen shoulder, its etiology is not known precisely. The clinical findings, course and prognosis are known with the researches. Although its incidence in the general population is %2-5, it is more likely to be seen in women between the ages of 40-70 and more than men. There are two types, primary and secondary. Primary frozen shoulder is idiopathic. Secondary frozen shoulder develops secondary to trauma, immobilization, rotator cuff tears, diabetes, biceps tendinitis, myocardial infarction, cerebrovascular event, psychological disorders, and post-surgical causes. Soft tissue contracture and adhesions in the capsule and axillary space are also seen in the pathogenesis. It is examined clinically in three stages. The first phase lasts about 0-3 months, when the intensity of the pain is high and the limitation of shoulder movements begins gradually. In the second stage, the severity of the pain slightly decreases, but the limitation of joint motion gradually increases, functionality decreases and lasts for about 3-9 months. In the third stage, the severity of the pain decreases, the joint movement limitations begin to recover slowly and gradually and lasts about 9-15 months. The treatment program shaped according to the characteristics of the stages; It includes conservative treatment approaches consisting of patient education, prevention, medical treatment, physiotherapy and exercises, and may require surgical treatment depending on the severity of the prognosis. Patient education in conservative treatment, hot packs, Transcutaneous Electrical Nerve Stimulation (TENS), Ultrasound (US), Laser, Iontophoresis etc. Electrotherapy agents, non-steroidal anti-inflammatory drugs (NSAIDs), corticosteroid injections, taping, joint and soft tissue mobilizations, manual therapy techniques and therapeutic exercises such as stretching exercises, range of motion exercises, proprioceptive neuromuscular facilitation techniques are frequently used.

Restriction in shoulder movements is quite evident especially in flexion, abduction and external rotation movements. Contracture of the ligaments in the shoulder reduces the volume of the capsule. The capsule decreasing in volume causes limitation of movement. However, the pain is not only due to the tension in the capsular and ligaments, but also due to the tension in the muscles and fascia and trigger toxins. Many therapeutic methods are used to relieve these trigger points and facial tensions. One of these methods is the "myofascial release technique" that focuses on soft tissues that are particularly tense and in spasm. This technique is a treatment method aimed at resolving fascial adhesions, restoring the optimal length of the muscle, reducing pain and increasing functionality.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with adhesive capsulitis
* Being 18 years or older
* Agree to voluntarily participate in research

Exclusion Criteria:

* Cervical disc hernias
* Neuromuscular diseases
* Full thickness rotator cuff tears
* Shoulder impingement syndrome
* Individuals with corticosteroid injection into the shoulder joint
* Individuals who have undergone surgical procedures on the shoulder joint
* Individuals with bone tumors or other malignant diseases
* Having mental and cognitive problems
* Physiotherapy or manual therapy on the same shoulder 6 months ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Change between baseline and first and 3 weeks
  Pain sensations are scored between 0 and 10. 0 is the lowest pain, 10 the highest pain.
Range of motion (ROM) with Goniometer | Change between baseline and first and 3 weeks
  Shoulder joint range of motion, The range of motion is measured between 0-180 degrees of flexion, 0-60 degrees of extension, 0-180 degrees of abduction, 0-50 degrees of abduction, internal rotation 0-90 degrees, external rotation 0-90 degrees.
Arm, Shoulder and Hand Problems Questionnaire (DASH) | Change between baseline and first and 3 weeks
  Upper extremity functionality levels, a value from 0 to 100 is obtained. The higher the score, the higher the degree of disability.
Shoulder Pain and Disability Index (SPADI) | Change between baseline and first and 3 weeks
  Specific shoulder pain and functions, all scores add up. The higher the score, the higher the degree of disability.
Pittsburgh Sleep Quality Index (PUKİ) | Change between baseline and first and 3 weeks
  Sleep quality, the scoring of the scale, which is evaluated by scoring each item between zero and three, is between 0-20. A total score higher than five indicates poor sleep quality.
Short Form-36 (SF-36) | Change between baseline and first and 3 weeks
  Quality of life, scoring of the scale is between 0-100. 100 is the highest score, 0 is the lowest.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Ataş Balcı, Assist Prof, Study Director — Bahçeşehir University
Locations (1):
- Private Levent Hospital, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No